CLINICAL TRIAL: NCT05102630
Title: The Use of Mechanical Ventilation Strategies and Its Potential Adverse Events Among ICU Patients With COVID-19 - a National-wide Retrospective Observational Study.
Brief Title: Ventilator Strategies in ICU Patients With COVID-19 - a National-wide Retrospective Observational Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Aalborg University Hospital (Other); Bispebjerg Hospital (Other); Herlev and Gentofte Hospital (Other); Hvidovre University Hospital (Other); Rigshospitalet, Denmark (Other); Aarhus University Hospital (Other); Region Zealand (Other)
Responsible Party: Principal Investigator, Anne Craveiro Brøchner, Ph D, associate professor, University of Southern Denmark
Other Study IDs: 2020-C 19-29-10-21
Record Dates: First submitted 2021-10-29; First posted 2021-11-01 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: ARDS Due to COVID-19
Keywords: ARDS; Mechanical Ventilation; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mechanical ventilation is likely lifesaving in patients with coronavirus disease 2019 (COVID-19) but may also result in adverse events. Only few studies describe the strategies used and adverse effect of mechanical ventilation in an unselected population of ICU patients with COVID-19.

This study is designed to be a retrospective study focusing on all mechanical ventilated ICU patients with COVID-19 included in the national Danish COVID ICU database between 10.03.2020 - 02.04.2021 i.e. a total of 1,193 patients. The investigators will register the use of the core interventions around mechanical ventilation and its potential adverse event, including barotrauma and prolonged ventilation.

This study will provide important data on the ventilation strategies used and its potential adverse events in unselected ICU patients with COVID-19 and thereby inform clinicians, patients, policy-makers, and future research in this area.

ELIGIBILITY:
Inclusion Criteria:

All mechanical ventilated patients registered in the national Danish COVID ICU database between 10.03.2020 - 02.04.2021 i.e.

1. Admitted to an ICU in Denmark
2. Laboratory-confirmed SARS-CoV-2 infection
3. Use of invasive mechanical ventilation (ventilation via a cuffed endotracheal tube) at any time during the ICU stay

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All mechanical ventilated patients registered in the national Danish COVID ICU database
Sampling Method: Probability Sample
Enrollment: 1193 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Ventilator days with lung -protective ventilation in percent of all ventilation days with 95%-CI. | Until 90 days
  Low tidal volume ventilation (Vt 4-8 mL/kg of predicted body weight)

SECONDARY OUTCOMES:
Pneumothorax | Until 90 days
  Pneumothorax noted in the medical record
Ventilator days | Until 90 days
  Number of days where the patients where the patient is ventilator depended
Number of patients with prolonged ventilation | Until 90 days
  Patients with more than 30 ventilator days
paO2/FiO2 ratio on days of ventilation | Until 90 days
  Ratio between measured arterial oxygen pressure and the fraction of inhaled oxygen
The use of APRV | Until 90 days
  The use of Airway pressure release as primary ventilator setting
Prone position | Until 90 days
  The use of prone position within the first 3 days and the use of prone position after day 3
Time to spontaneous ventilation | Until 90 days
  Time measured in days until the patients no longer needs controlled ventilation
Tracheostomy | Until 90 days
  Day after first intubation, Percutaneous dilatational tracheostomy (y/n), Surgical tracheostomy (y/n)
Adjuvant drugs | Until 90 days
  Adjuvant drugs at any time during mechanical ventilation
Mortality | Until 90 days
  Mortality at day 90

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Brøchner, MD, PhD, Principal Investigator — University of Southern Denmark
Locations (2):
- Denmark (2):
  - Department of Anaesthesiology and Intensive Care Medicine, Aalborg University Hospital, Aalborg
  - Department of Anesthesiology and Intensive Care, Kolding Hospital, Kolding

IPD SHARING:
Plan to Share IPD: No